CLINICAL TRIAL: NCT05338632
Title: Reversal of Opioid-induced Respiratory Depression With Opioid Antagonists - a Study in Opioid naïve Individuals and Chronic Opioid Users Under Real-life Conditions
Brief Title: Reversal of Opioid-induced Respiratory Depression With Opioid Antagonists
Acronym: ROAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: U.S. Food and Drug Administration (FDA) (Unknown)
Responsible Party: Principal Investigator, Albert Dahan, Professor, Leiden University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P21.112
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Opioid Induced Respiratory Depression; Chronic Opioid Use
Keywords: Reversal of opioid induced respiratory depression; Intranasal naloxone
MeSH Terms: interventions — Naloxone; Nasal Sprays; nalmefene

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized (IM versus IN naloxone), crossover study in a mixed population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Intravenous fentanyl year 1 (Experimental): continuous intravenous infusion of fentanyl to induce 40-60% respiratory depression.
  Interventions: Drug: Narcan 40 MG/ML Nasal Spray
- Intravenous sufentanil year 1 (Experimental): continuous intravenous infusion of sufentanil to induce 40-60% respiratory depression.
  Interventions: Drug: Narcan 40 MG/ML Nasal Spray
- Intravenous fentanyl year 2 (Experimental): continuous intravenous infusion of fentanyl to induce 40-60% respiratory depression.
  Interventions: Drug: Naloxone Hydrochloride; Drug: Nalmefene HCl injection
- IV fentanyl year 2 (Experimental): continuous intravenous infusion of fentanyl to induce 40-60% respiratory depression.
  Interventions: Drug: Naloxone Hydrochloride; Drug: Nalmefene HCl injection

INTERVENTIONS:
Drug: Narcan 40 MG/ML Nasal Spray — naloxone 4mg/0.1 mL intranasal spray, up to 4 doses intranasally, followed by 1ml 0.4 mg/ml naloxone hydrochloride intravenously
  Other Names: Intranasal naloxone
  Arms: Intravenous fentanyl year 1; Intravenous sufentanil year 1
Drug: Naloxone Hydrochloride — Naloxone 0.4mg/mL
  Other Names: IV naloxone
  Arms: IV fentanyl year 2; Intravenous fentanyl year 2
Drug: Nalmefene HCl injection — Nalmefene 1 ng/mL
  Other Names: Nalmefene IV
  Arms: IV fentanyl year 2; Intravenous fentanyl year 2

SUMMARY:
n this pharmacokinetic/pharmacodynamic modelling study we will determine the ability of intranasal and intravenous naloxone and intravenous nalmefene to reverse opioid (fentanyl and sufentanil)- induced respiratory depression in healthy volunteers and chronic opioid users to develop dosing recommendations in case of opioid-induced respiratory depression from an opioid overdose in clinical practice and in the out-of-hospital overdose.

DETAILED DESCRIPTION:
Primary objective:

To describe the pharmacokinetics and pharmacodynamics of intravenous fentanyl and sufentanil on ventilation of intranasal and intravenous naloxone and intravenous nalmefene in its ability to reverse respiratory depression (important model parameters include C50, a measure of potency and t½ke0). The results of these studies will allow us to perform simulation studies aimed at optimizing dosing regimens for intranasal and intramuscular naloxone in individuals that overdosed on potent opioids, with respiratory depression ranging from moderate to severe.

Secondary objectives:

To describe the pharmacokinetics and pharmacodynamics of intravenous fentanyl and sufentanil on pupil diameter and intranasal and intravenous naloxone and intravenous nalmefene in its ability to reverse miosis (important model parameters include C50, a measure of potency and t½ke0). The results of these studies will allow us to compare the ventilatory and pupil effects of the opioids and of naloxone.

Study design:

This is an open-label, randomized, crossover study in a mixed population

Study population:

We will study 12 healthy individuals of either sex aged 18-55 years and 12 individuals that are chronic opioids users (> 60 daily oral morphine equivalents; 18-55 years).

Intervention:

Study 1: Infusion of low-dose fentanyl and sufentanil whilst measuring minute ventilation and pupil diameter. When ventilation has dropped by 40-60% (Saturation > 85%), intranasal naloxone (IN, 4 mg) will be administered twice with a maximum of 180 minutes in between. At the end of each experiment 0.4 mg naloxone will be administered intravenously to determine its effect on ventilation and to allow calculation of naloxone intranasal bioavailability.

Study 2: Infusion of low-dose fentanyl whilst measuring minute ventilation and pupil diameter. When ventilation has dropped by 40-60% (Saturation > 85%), intravenous naloxone (IV, 0.4mg/mL) or intravenous nalmefene (IV, 1 mg/mL) will be administered at 5 min intervals with each bolus is 0.08 mg.

At regular intervals blood will be drawn for measurement of drug concentration; at regular intervals pupil diameter will be measured.

Main study parameters:

The main study measurement is minute ventilation. Together with the plasma concentration of the opioid and naloxone and nalmefene), ventilation is inputted in the PKPD model to get meaningful model parameters such as C50 and t½ke0, measures of potency and the speed of onset/offset of effect, respectively.

The secondary study measurement is pupil diameter. Together with the plasma concentration of the opioid and naloxone and nalmefene), the pupil diameter is inputted in the PKPD model to get meaningful model parameters such as C50 and t½ke0, measures of potency and the speed of onset/offset of effect, respectively. See Data analysis below. Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

In this pharmacokinetic-pharmacodynamic modeling study, the effect of intravenous and intranasal naloxone and intravenous nalmefene is studied during infusion of two opioids, fentanyl and sufentanil, in mixed population of healthy volunteers and chronic opioid users. The PK/PD analysis will yield important information regarding dosing regimens of IM and IN naloxone at fentanyl and sufentanil doses much higher than we will administer here, but that may represent doses in case of an overdose both in clinical patients and opioid abusers. Side effects related to the medication will be mild to moderate with most common side effects: nausea, vomiting, dizziness, somnolence, dry mouth and respiratory depression (from the opioids), and possibly mild withdrawal symptoms from naloxone. Side effects will dissipate over time while severe occurrences of nausea and vomiting will be treated with an antiemetic; severe occurrence of withdrawal symptoms will be treated with clonidine.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

1. Signed the informed consent form (ICF) and able to comply with the study requirements and restrictions listed therein;
2. Male and female subjects, age 18 to 70 years, inclusive;
3. Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have a negative serum pregnancy test prior to enrolment and must agree to use a medically acceptable means of contraception from screening through at least 1 month after the last dose of study drug;
4. Body Mass Index (BMI) 18 to 30 kg/m2, inclusive;
5. Healthy as defined by the Investigator, based on a medical evaluation that includes the subject's medical and surgical history, physical examination, vital signs, lab chemistry: estimated glomerular filtration rate >60 mL/min as estimated by the CKD-EPI equation, and AST or ALT levels < 3.0 times the upper limit of normal at screening, and negative serology tests for HIV, acute hepatitis B, or acute hepatitis C;
6. No history of substance use disorder;

Chronic opioid users

1. Signed the consent form and able to comply with the requirements and restrictions listed therein;
2. Males or females age 18 to 70 years, inclusive;
3. Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have a negative serum pregnancy test prior to enrolment and must agree to use a medically acceptable means of contraception from screening through at least 1 3 month after the last dose of study drug.
4. BMI 18 to 32 kg/m2, inclusive;
5. Opioid tolerant patients administered prescription opioids at daily doses ≥ 60 mg oral morphine equivalents (See Table 3);
6. Stable as defined by the Investigator, based on a medical evaluation that includes the subject's medical and surgical history, physical examination, vital signs, 12-lead ECG, hematology, and blood chemistry;

Exclusion Criteria:

Healthy volunteers

1. Currently meet the criteria for diagnosis of substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria on any substance;
2. Any other active medical condition, organ disease or concurrent medication or treatment that may either compromise subject safety or interfere with study endpoints;
3. Consume, on average, >27 20 units/week of alcohol in men and > 20 13 units/week of alcohol in women (1 unit = 1 glass (250 mL) beer, 125 mL glass of wine or 25 mL of 40% spirit);
4. Previous or current treatment with opioid agonist, partial agonist, or antagonist treatment within 30 days prior to the first study drug administration;
5. Significant traumatic injury, major surgery, or open biopsy within the prior 4 weeks of informed consent;
6. History of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent;
7. Measured systolic blood pressure greater than 160 or less than 95 mmHg or diastolic pressure greater than 95 mmHg at screening;
8. History or presence of allergic response to fentanyl, sufentanil or naloxone;
9. Subjects who have demonstrated allergic reactions (e.g., food, drug, atopic reactions or asthmatic episodes) which, in the opinion of the Investigator and sponsor, interfere with their ability to participate in the trial;
10. Treatment with another investigational drug within 3 months prior to dosing or having participated in more than 4 investigational drug studies within 1 year prior to screening;
11. Site staff or subjects affiliated with, or a family member of, site staff directly involved in the study;

Chronic opioid users

1. Currently meet the criteria for diagnosis of moderate or severe substance use disorder according to the DSM-5 criteria on any substances other than opioids, caffeine, or nicotine;
2. Any active medical condition, organ disease or concurrent medication or treatment that may either compromise subject safety or interfere with study endpoints;
3. Consume, on average, >27 units/week of alcohol in men and >20 units/week of alcohol in women (1 unit = 1 glass (250 mL) beer, 125 mL glass of wine or 25 mL of 40% spirit);
4. Currently receiving medication-assisted treatment for the treatment of opioid-use disorder;
5. Significant traumatic injury, major surgery, or open biopsy within the prior 4 weeks of informed consent;
6. History of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent;
7. Measured systolic blood pressure greater than 160 or less than 95 mmHg or diastolic pressure greater than 95 mmHg at screening;
8. History or presence of allergic response to study medication;
9. Opioid tolerant patients who have demonstrated allergic reactions (e.g., food, drug, atopic reactions or asthmatic episodes) which, in the opinion of the Investigator and sponsor, interfere with their ability to participate in the trial.
10. Estimated glomerular filtration rate <60 mL/min as estimated by the CKD-EPI equation;
11. Anemia at screening or donation of > 250 mL of blood or plasma within the last 3 months;
12. Positive serology tests for HIV, acute hepatitis B, or acute hepatitis C (OT patients with asymptomatic hepatitis B or C infection may be enrolled);
13. AST or ALT levels >3.0 times the upper limit of normal at screening;
14. Treatment with another investigational drug within 3 months prior to dosing or having participated in more than 4 investigational drug studies within 1 year prior to screening;
15. Site staff or subjects affiliated with, or a family member of, site staff directly involved in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Minute ventilation | Minute ventilation will be measured for up to 180 minutes following the start of opioid infusion
  Minute ventilation (liters/minute)
Plasma concentration sufentanil/fentanyl | at 2,5,10,15,20 and 30 minutes following opioid infusion and following every administration of intranasal/intravenous naloxone or nalmefene
  50 samples of 2ml arterial blood
Plasma concentration naloxone | at 2,5,10,15,20 and 30 minutes following opioid infusion and following every administration of intranasal/intravenous naloxone or nalmefene
  50 samples of 2ml arterial blood

SECONDARY OUTCOMES:
Pupil diameter | at 2,5,10,15,20 and 30 minutes following opioid infusion and following every administration of intranasal/intramuscular/intravenous naloxone. After discontinuation of infusion every 20 min. up to 6 hrs. following the start of opioid infusion
  Pupil diameter in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Rutger van der Schrier, MD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (texts, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed at. A.Dahan@lumc.nl

REFERENCES:
- [Background] Algera MH, Kamp J, van der Schrier R, van Velzen M, Niesters M, Aarts L, Dahan A, Olofsen E. Opioid-induced respiratory depression in humans: a review of pharmacokinetic-pharmacodynamic modelling of reversal. Br J Anaesth. 2019 Jun;122(6):e168-e179. doi: 10.1016/j.bja.2018.12.023. Epub 2019 Feb 1. PMID 30915997
- [Background] Algera MH, Olofsen E, Moss L, Dobbins RL, Niesters M, van Velzen M, Groeneveld GJ, Heuberger J, Laffont CM, Dahan A. Tolerance to Opioid-Induced Respiratory Depression in Chronic High-Dose Opioid Users: A Model-Based Comparison With Opioid-Naive Individuals. Clin Pharmacol Ther. 2021 Mar;109(3):637-645. doi: 10.1002/cpt.2027. Epub 2020 Oct 5. PMID 32865832
- [Background] Dahan A, Aarts L, Smith TW. Incidence, Reversal, and Prevention of Opioid-induced Respiratory Depression. Anesthesiology. 2010 Jan;112(1):226-38. doi: 10.1097/ALN.0b013e3181c38c25. PMID 20010421
- [Background] Olofsen E, van Dorp E, Teppema L, Aarts L, Smith TW, Dahan A, Sarton E. Naloxone reversal of morphine- and morphine-6-glucuronide-induced respiratory depression in healthy volunteers: a mechanism-based pharmacokinetic-pharmacodynamic modeling study. Anesthesiology. 2010 Jun;112(6):1417-27. doi: 10.1097/ALN.0b013e3181d5e29d. PMID 20461002
- [Background] Olofsen E, Boom M, Nieuwenhuijs D, Sarton E, Teppema L, Aarts L, Dahan A. Modeling the non-steady state respiratory effects of remifentanil in awake and propofol-sedated healthy volunteers. Anesthesiology. 2010 Jun;112(6):1382-95. doi: 10.1097/ALN.0b013e3181d69087. PMID 20461001
- [Background] van Dorp E, Yassen A, Dahan A. Naloxone treatment in opioid addiction: the risks and benefits. Expert Opin Drug Saf. 2007 Mar;6(2):125-32. doi: 10.1517/14740338.6.2.125. PMID 17367258
- [Background] Yassen A, Olofsen E, van Dorp E, Sarton E, Teppema L, Danhof M, Dahan A. Mechanism-based pharmacokinetic-pharmacodynamic modelling of the reversal of buprenorphine-induced respiratory depression by naloxone : a study in healthy volunteers. Clin Pharmacokinet. 2007;46(11):965-80. doi: 10.2165/00003088-200746110-00004. PMID 17922561
- [Background] Gepts E, Shafer SL, Camu F, Stanski DR, Woestenborghs R, Van Peer A, Heykants JJ. Linearity of pharmacokinetics and model estimation of sufentanil. Anesthesiology. 1995 Dec;83(6):1194-204. doi: 10.1097/00000542-199512000-00010. PMID 8533912